# Imperial College London

Research Governance and Integrity Team



Intra-operative Ultrasound Guided Ovarian Cystectomy as a Method of Fertility Preservation (UGLOC): A Randomised Controlled Trial

Date: 15/06/2021

IRAS Number: 290747

### Imperial College London

Research Governance and Integrity Team



Please initial hox

#### **Informed Consent Form**

DOCUMAS: 20QC6370

#### **Full Title of Project:**

Intra-operative ultrasound guided laparoscopic ovarian cystectomy (UGLOC) as a method of fertility preservation in the management of benign ovarian cysts: A Randomised Controlled Trial.

Name of Principal Investigator: Mr Joseph Yazbek

| | | 1 icuse | IIII DOA |
|---|---|---|---|
| 1. | I confirm that I have read and understand the participant information sheet dated 30.7.21 version 6 or the above study and have had the opportunity to ask questions which have been answered fully. | | |
| 2. | I understand that my participation is voluntary and I am free to withdraw at any time, without giving any reason and without my medical care or legal rights being affected. | | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from the research group from Imperial College London, NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. | | |
| 4. | I give permission for these individuals to access my records that are relevant to this research. | | |
| 5. | I consent for information collected about me to be used to support other research in the future, including those outside of the EEA. (Circle as appropriate Yes/No) | Yes [/No | |
| 6. | I give permission for members of the research team to contact my GP with details of my participation in the study and the post-operative follow up findings. | | |
| 7. | I consent to take part in the above study. | | |
| 8. | I consent to being contacted to potentially taking part in other research studies. (Circle as appropriate Yes/No) | Yes [ | |

IRAS No: 290747 V4.0 15 June 2021 Page 2 of 3

# Imperial College London

### Research Governance and Integrity Team



| | | Please initial box |
|---|---|---|
| 9. I consent to being contacted at th results obtained from the study (Cir | • | · — |
| | | Yes<br>/No |
| Name of Subject | Signature | Date |
| Name of Person taking consent | Signature | Date |

 $1\ copy\ for\ Subject;\ 1\ copy\ for\ Principal\ Investigator;\ 1\ copy\ to\ be\ kept\ with\ hospital\ notes$